CLINICAL TRIAL: NCT00470236
Title: A Randomised Phase III Study of Radiation Doses and Fractionation Schedules in Non-low Risk Ductal Carcinoma In Situ (DCIS) of the Breast
Brief Title: Radiation Doses and Fractionation Schedules in Non-low Risk Ductal Carcinoma In Situ (DCIS) of the Breast
Acronym: DCIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Breast International Group (Other); NCIC Clinical Trials Group (Network); Cancer Trials Ireland (Network); Borstkanker Onderzoek Groep (Network); ETOP IBCSG Partners Foundation (Network); Scottish Cancer Trials Breast Group (Unknown); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 07.01; NHMRC 454390 (Other Grant/Funding Number: NHMRC); BIG 3-07 (Other: Collaborative Group); NCIC CTG MA.33 (Other: Collaborative Group); BOOG 2009-03 (Other: Collaborative Group); ICORG 10-06 (Other: Collaborative Group); EORTC 22085-10083 (Other: Collaborative Group); IBCSG 38-10 (Other: Collaborative Group); SCTBG 2009MayPR55 (Other: Collaborative Group)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Ductal, Breast
Keywords: Ductal carcinoma in-situ; Breast conserving therapy; Whole breast radiation therapy; Tumour bed boost; Fractionation schedules; Completely excised non-low risk DCIS
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Carcinoma, Intraductal, Noninfiltrating | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Standard WB Fractionation) (Active Comparator): Whole Breast RT alone - Standard fractionation schedule (50GY/25 Fractions/35days)
  Interventions: Radiation: Standard WB fractionation
- Arm 2 (Shorter WB Fractionation) (Experimental): Whole Breast RT alone - Shorter fractionation schedule (42.5 Gy/16 fractions/22 days)
  Interventions: Radiation: Shorter WB fractionation
- Arm 3 (Standard WB fractionation+Boost) (Active Comparator): Whole Breast RT + tumor bed boost - Standard fractionation schedule (50 Gy/25 fractions/35 days; Boost 16 Gy/8 fractions/10 days)
  Interventions: Radiation: Standard WB fractionation+Boost
- Arm 4 (Shorter WB fractionation + Boost) (Experimental): Whole breast RT + tumour bed boost - Shorter fractionation schedule (42.5 Gy/16 fractions/22 days; Boost 16 Gy/8 fractions/10 days)
  Interventions: Radiation: Shorter WB fractionation + Boost

INTERVENTIONS:
Radiation: Standard WB fractionation — A total dose of 50 Gy in 25 fractions in 2-Gy daily fractions, 5 fractions per week (at least 9 fractions per fortnight).
  Other Names: Radiation
  Arms: Arm 1 (Standard WB Fractionation)
Radiation: Shorter WB fractionation — A total dose of 42.5 Gy in 16 fractions in 2.656-Gy daily fractions, 5 fractions per week (at least 9 fractions per fortnight).
  Other Names: Radiation
  Arms: Arm 2 (Shorter WB Fractionation)
Radiation: Standard WB fractionation+Boost — Whole Breast: A total dose of 50 Gy in 25 fractions in 2-Gy daily fractions, 5 fractions per week (at least 9 fractions per fortnight).
  Tumour bed: A total dose of 10 Gy in 5 fractions in 2-Gy daily fractions, 5 fractions per week.
  Other Names: Radiation
  Arms: Arm 3 (Standard WB fractionation+Boost)
Radiation: Shorter WB fractionation + Boost — Whole breast: A total dose of 42.5 Gy in 16 fractions in 2.656-Gy daily fractions, 5 fractions per week (at least 9 fractions per fortnight).
  Tumour bed: A total dose of 10 Gy in 4 fractions in 2.5-Gy daily fractions, 4 fractions per week.
  Other Names: Radiation
  Arms: Arm 4 (Shorter WB fractionation + Boost)

SUMMARY:
Hypotheses:

1. The addition of tumour bed boost after BCS in women with non-low risk DCIS reduces the risk of local recurrence (invasive or intraductal recurrence in the ipsilateral breast).
2. The risk of local recurrence in the shorter fractionation arm is not worse than that for the standard fractionation arm.
3. A molecular signature predictive of invasive recurrence of DCIS will be detectable and the molecular signature may eventually have clinical utility for therapy individualization.

Overall Objectives:

1. To improve the outcome of women with non-low risk DCIS treated with breast conserving therapy.
2. To individualize treatment selection for women with DCIS to achieve long term disease control with minimal toxicity.

DETAILED DESCRIPTION:
Specific objectives:

1. To evaluate time to local recurrence in women with DCIS treated with breast conserving surgery followed by:

   * whole breast RT alone versus whole breast RT plus tumour bed boost;
   * RT using the standard fractionation schedule versus the shorter schedule.
2. To evaluate time to disease recurrence and overall survival in women with DCIS treated with breast conserving surgery followed by:

   * whole breast RT alone versus whole breast RT plus tumour bed boost;
   * RT using the standard fractionation schedule versus the shorter schedule.
3. To compare the toxicity of:

   * whole breast RT alone versus whole breast RT plus tumour bed boost;
   * RT using the standard fractionation schedule versus the shorter schedule.
4. To compare the cosmetic outcome of:

   * whole breast RT alone versus whole breast RT plus tumour bed boost;
   * RT using the standard fractionation schedule versus the shorter schedule.
5. To identify a molecular signature predictive of invasive recurrence of DCIS to facilitate therapy individualization.
6. To assess inter-relationship of biomarkers and relationship between biomarker expression and specific histopathologic features of DCIS.
7. To evaluate the quality of life of women treated with:

   * whole breast RT alone versus whole breast RT plus tumour bed boost;
   * RT using the standard fractionation schedule versus the shorter schedule.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria for admission to study:

* Women ≥ 18 years.
* Histologically proven DCIS of the breast without an invasive component.
* Bilateral mammograms performed within 6 months prior to randomization.
* Clinically node-negative.
* Treated by breast conserving surgery (primary excision or re-excision) with complete microscopic excision and clear radial margins of ≥1 mm* (*Patients with superficial or deep resection margin of <1 mm are eligible if surgery has removed all of the intervening breast tissue from the subcutaneous tissue to the pectoralis fascia).
* Women who are at high risk of local recurrence due to:

  * Age < 50 years; OR
  * Age ≥ 50 years plus at least one of the following:

    * Symptomatic presentation
    * Palpable tumour
    * Multifocal disease
    * Microscopic tumour size ≥ 1.5 cm in maximum dimension
    * Intermediate or high nuclear grade
    * Central necrosis
    * Comedo histology
    * Radial* surgical resection margin < 10 mm. (*Patients with superficial or deep resection margin of < 10 mm are eligible if surgery has not removed all of the intervening breast tissue from the subcutaneous tissue to the pectoralis fascia.)
* Assessed by surgeon and radiation oncologist to be suitable for breast conserving therapy including whole breast RT.
* Ability to tolerate protocol treatment.
* Protocol RT should preferably commence within 8 weeks but must commence no later than 12 weeks from the last surgical procedure.
* ECOG performance status 0, 1 or 2.
* Patient's life expectancy > 5 years.
* Availability for long-term follow-up.
* Written informed consent.

Exclusion Criteria:

Patients who fulfill any of the following criteria are not eligible for admission to study:

* Multicentric disease or extensive microcalcifications that could not be completely excised by breast conserving surgery with radial margins of ≥1 mm*.

  *Patients with superficial and/or deep margin of <1 mm are eligible if surgery has removed all of the intervening breast tissue from the subcutaneous tissue to the pectoralis fascia.
* Presence of tumour cells in lymph nodes detected using H&E or immunohistochemical examination (if lymph node biopsy or dissection has been performed).
* Locally recurrent breast cancer.
* Previous DCIS or invasive cancer of the contralateral breast.

  * Bilateral DCIS of the breasts
  * Synchronous invasive carcinoma of the contralateral breast
* Other concurrent or previous malignancies except:

  * Non-melanomatous skin cancer;
  * Carcinoma in situ of the cervix or endometrium; and
  * Invasive carcinoma of the cervix, endometrium, colon, thyroid and melanoma treated at least five years prior to study admission without disease recurrence.
* Serious non-malignant disease that precludes definitive surgical or radiation treatment (e.g., scleroderma, systemic lupus erythematosus, cardiovascular/pulmonary/renal disease).
* ECOG performance status ≥ 3.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1608 (Actual)
Dates: Start 2007-06; Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Time to local recurrence, measured from the date of randomization to the date of first evidence of local recurrence. | Main analysis after all patients have completed 5 years of follow-up. Updated analysis after 10 years of follow-up.

SECONDARY OUTCOMES:
Overall survival | Measured from the date of randomization to the date of death from any cause. Main analysis of secondary outcomes after all patients have completed 5 years of follow-up. Updated analysis after 10 years of follow-up.
Time to disease recurrence | Measured from the date of randomization to the date of first evidence of recurrent disease. Main analysis of secondary outcomes after all patients have completed 5 years of follow-up. Updated analysis after 10 years of follow-up.
Cosmetic Outcome | Cosmetic assessment will take place at baseline, 12, 36 and 60 months post RT.
Radiation toxicity | Assessed at baseline, last week of RT, 3, 6, and 12 months post RT and then yearly until year 10.
Quality of Life change | Assessed at baseline, last week of RT, 6, 12, 24, 60 & 120 months post RT.

CONTACTS AND LOCATIONS:
Overall Officials: Boon Chua, Study Chair — Prince of Wales Hospital Randwick
Locations (120):
- Australia (26):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Nepean Cancer Care Centre, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Premion - Wesley, Auchenflower, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Genesis Cancer Care (previously Premion) - Nambour, Nambour, Queensland
  - Radiation Oncology - Mater Centre, South Brisbane, Queensland
  - Toowoomba Cancer Research Centre, Toowoomba, Queensland
  - North Queensland Oncology Service, Townsville, Queensland
  - Genesis Cancer Care (previously Premion) - Tugun, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Barwon Health - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - William Buckland Radiotherapy Centre, Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gardiner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Perth Radiation Oncology, Perth, Western Australia
- Belgium (7):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - ZNA Middelheim, Antwerp
  - Cliniques Univeritaires St Luc, Brussels
  - Universitair Zielenhusi, Brussels
  - Hopital De Jolimont, Haine-Saint-Paul
  - AZ Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - Algemeen Ziekenhis Sint-Augustinus, Wilrijk
- Canada (20):
  - Nova Scotia Cancer Centre, Halifax
  - Jurvanski Cancer Centre, Hamilton
  - Notre Dame Hospital, Hearst
  - BCCA Southern Interior - CAVK, Kelowna
  - London Regional Cancer Program, London
  - Saint John Regional Hospital, Miramichi
  - Leon Richard Oncology Centre, Moncton
  - Hospital Maisonneuve-Rosemont, Montreal
  - Lakeridge Health, Oshawa
  - CHUQ L'Hotel-Dieu de Quebec, Québec
  - McGill University Department of Oncology, Sainte-Anne-de-Bellevue
  - Allan Blair Cancer Centre, Saskatoon
  - Saskatoon Cancer Centre, Saskatoon
  - Universite de Sherbrooke - CUGH, Sherbrooke
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay
  - Odette Cancer Centre, Toronto
  - Princess Margaret Hospital, Toronto
  - BCCA Vancouver Centre, Victoria
  - Vancouver Island Cancer Centre, Victoria
  - Cancer Care Manitoba, Winnipeg
- France (2):
  - Chr De Grenoble - La Tronche, Grenoble
  - Centre Antine Lacassagne, Nice
- Ireland (3):
  - Cork University Hospital, Cork
  - University Hospital Galway, Galway
  - SLRON (St Luke's Rad Onc Network), Rathgar
- Italy (2):
  - Centro Di Riferimento Oncologico - Aviano, Aviano
  - Fondazione Salvatore Maugeri, Pavia
- Netherlands (9):
  - Academisch Medisch Centrum, Amsterdam
  - Cancer Institute Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Arnhem 'S Radiotherapeutisch Instituut, Arnhem
  - Reinier de Graaf Groep, Delft
  - University Medical Centre Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Maastricht Radiation Oncology Maastro Clinic, Maastricht
  - Medisch Centrum Haaglanden, Westeinde
  - ISALA Klinieken, Zwolle
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- National University Hospital, Singapore, Singapore
- Switzerland (8):
  - University Hospital Basel, Basel
  - IOSI, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubunden, Chur
  - Kantonsspital Munsterlingen, Münsterlingen
  - Kantonsspital St. Gallen, Sankt Gallen
  - Brust-Zentrum Zurich-Seefeld, Zurich
  - Klinik Hirslanden, Zurich
- United Kingdom (39):
  - Gloucestershire Royal & Cheltenham General Hospitals, Cheltenham, Gloucestershire
  - Churchill Hospital, Oxford, Headington
  - Pilgram Hospital, Boston, Lincolnshire
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Ealing Hospital, Southall, Middlesex
  - Kings Mill Hospital Nottingham, Sutton in Ashfield, Nottinghamshire
  - Musgrove Park Hospital, Taunton, Somerset
  - Queens Hospital Burton, Burton-on-Trent, Staffordshire
  - University of North Staffordshire, Stoke-on-Trent, Staffordshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Basildon University Hospital, Basildon
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Sandwell and West Birmingham Hospitals NHS Trust, Birmingham
  - Bristol Haematology & Oncology, Bristol
  - Colchester Hospital, Colchester
  - Coventry Arden Cancer Centre, Coventry
  - Royal Derby Hospital, Derby
  - Dumfries & Galloway Royal Infirmary, Dumfries
  - Queen Margaret Hospital, Dunfermline
  - Edinburgh Western General Hospital, Edinburgh
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Ipswich Hospital, Ipswich
  - Kidderminster Hospital, Kidderminster
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Imperial College Healthcare Charing Cross, London
  - James Cook University Hospital, Middlesbrough
  - Nottingham University Hospitals, Nottingham
  - Royal Alexandra Hospital, Paisley
  - Alexandra Hospital, Redditch
  - Weston Park Hospital, Sheffield
  - The Shrewsbury and Telford Hospital NHS Trust, Shrewsbury
  - Southend University Hopstial, Southend
  - Stafford Hospital, Stafford
  - Royal Marsden, Sutton
  - Warwick Hospital, Warwick
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Chua BH, Link EK, Kunkler IH, Whelan TJ, Westenberg AH, Gruber G, Bryant G, Ahern V, Purohit K, Graham PH, Akra M, McArdle O, O'Brien P, Harvey JA, Kirkove C, Maduro JH, Campbell ID, Delaney GP, Martin JD, Vu TTT, Muanza TM, Neal A, Olivotto IA; BIG 3-07/TROG 07.01 trial investigators. Radiation doses and fractionation schedules in non-low-risk ductal carcinoma in situ in the breast (BIG 3-07/TROG 07.01): a randomised, factorial, multicentre, open-label, phase 3 study. Lancet. 2022 Aug 6;400(10350):431-440. doi: 10.1016/S0140-6736(22)01246-6. PMID 35934006
- [Derived] King MT, Link EK, Whelan TJ, Olivotto IA, Kunkler I, Westenberg AH, Gruber G, Schofield P, Chua BH; BIG 3-07/TROG 07.01 trial investigators. Quality of life after breast-conserving therapy and adjuvant radiotherapy for non-low-risk ductal carcinoma in situ (BIG 3-07/TROG 07.01): 2-year results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2020 May;21(5):685-698. doi: 10.1016/S1470-2045(20)30085-1. Epub 2020 Mar 20. PMID 32203696
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au